CLINICAL TRIAL: NCT01453556
Title: Intracorporeal Versus Extracorporeal Mechanical Anastomosis in Laparoscopic Right Colectomy. A Prospective Randomized Controlled Clinical Trial
Brief Title: Intracorporeal Versus Extracorporeal Mechanical Anastomosis in Laparoscopic Right Colectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Scientific Institute San Raffaele (Other)
Responsible Party: Principal Investigator, Andrea Vignali, Principal Investigator, Scientific Institute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Intraextra01
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Last update posted 2011-10-21 (Estimated); Status verified 2011-10

CONDITIONS: Neoplastic or Benign Disease of Right Colon; Elective Laparoscopic Surgery
Keywords: Laparoscopic surgery; Right colectomy; Mechanical anastomosis; Post-operative ileum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intracorpopreal anastomosis (Experimental): Intracorporeal mechanical anastomosis
  Interventions: Procedure: Laparoscopic right colectomy
- Extracorporeal anastomosis (Active Comparator): Extracorporeal mechanical anastomosis
  Interventions: Procedure: Laparoscopic right colectomy

INTERVENTIONS:
Procedure: Laparoscopic right colectomy — Laparoscopic right colectomy with mechanical ileo-colon anastomosis L-L

SUMMARY:
Verify with a prospective randomised trial if intracorporeal mechanical anastomosis in laparoscopic right colectomy reduces post-operative bowel canalisation time and length of stay in comparison with extracorporeal mechanical anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or more
* Benign o neoplastic disease of right colon
* Elective laparoscopic surgery

Exclusion Criteria:

* Emergency surgery
* Adhesion or infiltration of near organs
* Severe heart disease ( New York Heart Association class > 3 )
* Severe respiratory disease ( arterial PO2 < 70 torr )
* Severe Liver disease (Child-Pugh class C)
* Ongoing infections
* Number of plasmatic neutrophil < a 2.0 x 10 9/L
* Other contraindications to laparoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Post-operative canalisation time and length of stay | Post-operative stay (about 7 days)
  Comparison of post-operative bowel movement time (fist flastus and first dejection) and overall length of stay between the two study groups

SECONDARY OUTCOMES:
Impact of post-operative ileum and complications. Valuation of global costs | 12 months
  Comparison of post-operative short and long-term complications (in particular post-operative ileum) between the two study groups. Valuation of global costs differences.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Vignali, MD, Principal Investigator — San Raffaele Scientific Institute; Carlo Staudacher, Prof, Study Director — San Raffaele Scientific Institute
Locations (1):
- San Raffaele Scientific Institute, Milan, MI, Italy